CLINICAL TRIAL: NCT00727038
Title: Randomized Controlled Trial of Lucentis in the Management of New Onset Neovascular Glaucoma
Brief Title: Lucentis for New Onset Neovascular Glaucoma
Acronym: NVG
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company withdrew funding/sponsorship
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Blair, Faculty Ophthalmology and Visual Services, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0792; FVF4143S (Other: Genentech, Inc.)
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2008-07

CONDITIONS: Glaucoma; New Onset Glaucoma; Neovascular Glaucoma; New Onset Neovascular Glaucoma
Keywords: glaucoma; neovascular glaucoma; new onset glaucoma; retinal ischemia; central retinal vein occlusion; proliferative diabetic retinopathy; ocular ischemic syndrome; carotid stenosis; vascular endothelial growth factor; neovascular
MeSH Terms: conditions — Glaucoma; Glaucoma, Neovascular; Retinal Vein Occlusion; Carotid Stenosis | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lucentis (ranibizumab) with conventional treatment
  Interventions: Drug: Ranibizumab (Lucentis)
- 2 (No Intervention): Conventional treatment

INTERVENTIONS:
Drug: Ranibizumab (Lucentis) — 0.5 mg ranibizumab intravitreal injection single dose administration
  Other Names: ranibizumab; Lucentis
  Arms: 1

SUMMARY:
Neovascular glaucoma is a potentially debilitating disease of the eye. Vascular eye disease such as diabetes and vein occlusions can cause the retina to release factors that promote the growth of abnormal blood vessels. These abnormal vessels can grow in the drainage mechanism of the eye causing pressure in the eye to markedly increase. This can potentially cause irreversible damage to the optic nerve from glaucoma leading to permanent blindness and painful eyes. Conventional treatments including laser and freezing therapy take weeks to cause regression in abnormal blood vessel growth. This delay often results in permanent vision loss and pain. New medications targeted at more immediately reducing blood vessel growth may aid in the treatment of this disease.

DETAILED DESCRIPTION:
Hypothesis:

Intravitreal injection of Lucentis prior to conventional treatment for neovascular glaucoma improves overall outcome compared to conventional treatment alone.

Specific Aims:

To determine if pre-treatment with a single intravitreal injection of Lucentis prior to conventional treatment prevents severe vision loss and improves intraocular pressure control compared to conventional treatment alone.

Neovascular glaucoma is a potentially devastating consequence of fibrovascular proliferation of the anterior chamber angle with subsequent obstruction of the trabecular meshwork. The production of peripheral anterior synechiae along the trabecular meshwork leads to progressive angle closure. The subsequent elevation in intraocular pressure is difficult to manage, often leading to rapid progression of glaucoma and significant loss of vision. Enucleation for blind, painful eyes secondary to neovascular glaucoma is not an uncommon sequelae.

Neovascular glaucoma has many etiologic causes, the vast majority resulting from retinal ischemia secondary to relatively common diseases such as central retinal vein occlusion, proliferative diabetic retinopathy and ocular ischemic syndrome (carotid stenosis). (Sivac-Callcott et al., 2001) Vascular endothelial growth factor is likely a major contributor to the development of angle and iris neovascularization. (Ferrara, 2004) Although panretinal photocoagulation and/or cryoablation are mainstays of conventional treatment for neovascular glaucoma, the delayed therapeutic effect of these interventions often results in the formation of peripheral anterior synechiae and permanent angle closure.

Recent limited case series have demonstrated a role for bevacizumab (Avastin) in reducing rubeosis iridis and as an adjunct for neovascular glaucoma. (Grisanti et al., 2006; Davidorf et al., 2006; Iliev et al., 2006; Kahook, Schuman, Noecker, 2006) However, no prospective studies have examined the potential utility of anti-vascular endothelial growth factor agents in the treatment of neovascular glaucoma. Intravitreal Lucentis is the standard of care for the treatment of exudative macular degeneration. Pharmacologic agents such as Lucentis, which selectively inhibit vascular endothelial growth factor may provide an important therapeutic adjunct for the treatment of neovascular glaucoma by more immediately causing regression of angle neovascularization and thereby providing a window for permanent treatment with laser or cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 21 years
* Diagnosis of neovascular glaucoma (angle neovascularization with or without iris neovascularization and IOP > 21 mm Hg and > 5 mm Hg IOP compared to the fellow eye).
* Neovascular glaucoma secondary to retinal ischemia (central retinal vein occlusion, proliferative diabetic retinopathy, ocular ischemic syndrome, etc.)

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation or pre-menopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* > 270 degrees of closed trabecular meshwork (closure secondary to peripheral anterior synechiae)
* History of active inflammatory, infectious, or idiopathic keratitis precluding view of the anterior segment structures.
* Previous intravitreal injections of ranibizumab or bevacizumab in either eye.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01-04 (Actual); Primary Completion 2009-05-15 (Actual); Study Completion 2009-05-15 (Actual)

PRIMARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters from baseline to Month 6. | Baseline to Month 6.

SECONDARY OUTCOMES:
Percent change in angle neovascularization (measured in clock hours by gonioscopy). | Initial visit through Month 6
Percent change in permanent angle closure (clock hours of peripheral anterior synechiae by gonioscopy). | Initial visit through Month 6
Mean change in intraocular pressure measured by applanation tonometry. | Initial visit through Month 6
Percent change in iris neovascularization (measured both in clock hours by slit lamp exam and with iris angiography). | Initial visit through Month 6
Rates of severe vision loss (visual acuity <20/200, loss of 6 lines or more on ETDRS chart). | Initial Visit through Month 6
Number of intraocular pressure lowering medications needed to control intraocular pressure. | Initial Visit through Month 6
Mean change in optic nerve cupping. | Initial Visit through Month 6
Percent of patients requiring surgical glaucoma procedure to control intraocular pressure (trabeculectomy, seton, or ciliary body destruction). | Study duration
Percent of patients requiring pars plana vitrectomy with endolaser. | Study duration
Rates of endophthalmitis. | Study duration
Rates of rhegmatogenous retinal detachment. | Study duration
Final clock hours of permanent angle closure (clock hours of peripheral anterior synechiae by gonioscopy) | Month 6 visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Blair, MD, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Background] Avery RL. Regression of retinal and iris neovascularization after intravitreal bevacizumab (Avastin) treatment. Retina. 2006 Mar;26(3):352-4. doi: 10.1097/00006982-200603000-00016. No abstract available. PMID 16508438
- [Background] Davidorf FH, Mouser JG, Derick RJ. Rapid improvement of rubeosis iridis from a single bevacizumab (Avastin) injection. Retina. 2006 Mar;26(3):354-6. doi: 10.1097/00006982-200603000-00017. No abstract available. PMID 16508439
- [Background] Ferrara N. Vascular endothelial growth factor: basic science and clinical progress. Endocr Rev. 2004 Aug;25(4):581-611. doi: 10.1210/er.2003-0027. PMID 15294883
- [Background] Fung AE, Rosenfeld PJ, Reichel E. The International Intravitreal Bevacizumab Safety Survey: using the internet to assess drug safety worldwide. Br J Ophthalmol. 2006 Nov;90(11):1344-9. doi: 10.1136/bjo.2006.099598. Epub 2006 Jul 19. PMID 16854824
- [Background] Iliev ME, Domig D, Wolf-Schnurrbursch U, Wolf S, Sarra GM. Intravitreal bevacizumab (Avastin) in the treatment of neovascular glaucoma. Am J Ophthalmol. 2006 Dec;142(6):1054-6. doi: 10.1016/j.ajo.2006.06.066. Epub 2006 Aug 2. PMID 17157590
- [Background] Kahook MY, Schuman JS, Noecker RJ. Intravitreal bevacizumab in a patient with neovascular glaucoma. Ophthalmic Surg Lasers Imaging. 2006 Mar-Apr;37(2):144-6. PMID 16583637
- [Background] Sivak-Callcott JA, O'Day DM, Gass JD, Tsai JC. Evidence-based recommendations for the diagnosis and treatment of neovascular glaucoma. Ophthalmology. 2001 Oct;108(10):1767-76; quiz1777, 1800. doi: 10.1016/s0161-6420(01)00775-8. PMID 11581047
- [Background] Results of the Endophthalmitis Vitrectomy Study. A randomized trial of immediate vitrectomy and of intravenous antibiotics for the treatment of postoperative bacterial endophthalmitis. Endophthalmitis Vitrectomy Study Group. Arch Ophthalmol. 1995 Dec;113(12):1479-96. PMID 7487614
- See also: University of Illinois at Chicago Eye and Ear Infirmary homepage — http://www.uic.edu/com/eye/